CLINICAL TRIAL: NCT03553836
Title: Adjuvant Therapy With Pembrolizumab Versus Placebo in Resected High-risk Stage II Melanoma: A Randomized, Double-blind Phase 3 Study (KEYNOTE-716)
Brief Title: Safety and Efficacy of Pembrolizumab Compared to Placebo in Resected High-risk Stage II Melanoma (MK-3475-716/KEYNOTE-716)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-716; MK-3475-716 (Other: MSD); KEYNOTE-716 (Other: MSD); 205203 (Registry Identifier: JAPIC-CTI); 2022-501966-23 (Registry Identifier: EU CT Number); U1111-1282-6109 (Other: Universal Trial Number); 2018-000669-35 (EudraCT Number)
Record Dates: First submitted 2018-06-01; First posted 2018-06-12 (Actual); Results first posted 2022-06-24 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Melanoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1(PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and Investigators will be blinded in Part 1 and unblinded in Part 2, if done.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants receive 200 mg pembrolizumab (2 mg/kg for a maximum of 200 mg in pediatric participants) by intravenous (IV) infusion once every 3 weeks (Q3W; 21-day cycles) for up to 17 cycles (up to ~1 year) in Part 1. Participants who complete the initial treatment of 17 cycles of pembrolizumab and experience disease recurrence may be eligible for re-challenge with pembrolizumab at the same dose and schedule of 200 mg Q3W (21-day cycles) for up to 35 cycles (up to ~2 years) in Part 2.
  Interventions: Biological: Pembrolizumab
- Placebo (Placebo Comparator): Participants receive saline placebo by IV infusion Q3W (21-day cycles) for up to 17 cycles (up to ~1 year) in Part 1. Participants who complete the initial treatment of 17 cycles of placebo and experience disease recurrence may be eligible to switch over to pembrolizumab 200 mg Q3W (21-day cycles) for up to 35 cycles (up to ~2 years) in Part 2.
  Interventions: Biological: Pembrolizumab; Other: Placebo

INTERVENTIONS:
Biological: Pembrolizumab — Administered as an intravenous (IV) infusion every 3 weeks (Q3W)
  Other Names: KEYTRUDA®; MK-3475
Other: Placebo — Administered as an IV infusion every 3 weeks (Q3W)
  Arms: Placebo

SUMMARY:
This 2-part study will evaluate the safety and efficacy of pembrolizumab (MK-3475) compared to placebo in participants with surgically resected high-risk Stage II melanoma. Participants in Part 1 will receive either pembrolizumab or placebo in a double-blind design every 3 weeks (Q3W) for up to 17 cycles/~1 year (each cycle = 21 days). Participants who complete the initial treatment of 17 cycles of pembrolizumab in Part 1 and experience disease recurrence may be eligible for re-challenge with pembrolizumab at the same dose and schedule of 200 mg Q3W (21-day cycles) for up to 35 cycles (up to ~2 years) in Part 2 in an open label design. Participants who complete the initial treatment of placebo and experience disease recurrence may be eligible to switch over to pembrolizumab 200 mg Q3W (21-day cycles) for up to 35 cycles (up to ~2 years) in Part 2 in an open label design. The primary hypothesis of this study is that pembrolizumab increases recurrence-free survival (RFS) compared to placebo.

Per protocol, response/ progression or adverse events (AEs) during re-challenge/switch-over in Part 2 will not be counted towards the RFS outcome measure or safety outcome measures respectively.

ELIGIBILITY:
Inclusion:

* Has surgically resected and histologically/pathologically confirmed new diagnosis of Stage IIB or IIC cutaneous melanoma per American Joint Committee on Cancer (AJCC) 8th edition guidelines
* Has not been previously treated for melanoma beyond complete surgical resection
* Has ≤12 weeks between final surgical resection and randomization
* Has no evidence of metastatic disease on imaging as determined by investigator
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale or Lansky Play-Performance Scale (LPS) score ≥50 for participants ≤16 years old, or a Karnofsky Performance Scale (KPS) score ≥50 for participants >16 and <18 years old
* Has recovered adequately from toxicity and/or complications from surgery prior to study start
* Female participants must not be pregnant or breastfeeding, and must agree to use contraception during the treatment period and for at least 120 days after the last dose of study treatment if they are women of childbearing potential (WOCBP)

Exclusion:

* Has a known additional malignancy that is progressing or has required active antineoplastic therapy (including hormonal) within the past 5 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* WOCBP who has a positive urine pregnancy test within 72 hours prior to randomization. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Has received prior therapy with an anti-Programmed Cell Death Receptor 1 (PD-1), anti-Programmed Cell Death Receptor Ligand 1 (PD-L1) or anti-Programmed Cell Death Receptor Ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, CD137)
* Has received prior systemic anti-cancer therapy for melanoma including investigational agents
* Has received a live vaccine within 30 days prior to the first dose of study treatment
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Has severe hypersensitivity (≥Grade 3) to any excipients of pembrolizumab
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of hepatitis B (defined as hepatitis B surface antigen reactive) or known active hepatitis C virus (defined as hepatitis C virus ribonucleic acid [RNA] [qualitative] is detected) infection
* Has a history of active tuberculosis (Bacillus tuberculosis)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Has had an allogeneic tissue/solid organ transplant

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 976 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2033-10-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (159):
- United States (39):
  - University of Arizona Cancer Center ( Site 0121), Tucson, Arizona
  - UCSD Moores Cancer Center ( Site 0133), La Jolla, California
  - The Angeles Clinic and Research Institute ( Site 0029), Los Angeles, California
  - UCLA Hematology & Oncology ( Site 0130), Los Angeles, California
  - John Wayne Cancer Institute ( Site 0026), Santa Monica, California
  - University of Colorado Cancer Center ( Site 0027), Aurora, Colorado
  - Yale University ( Site 0035), New Haven, Connecticut
  - Mayo Clinic Florida ( Site 0024), Jacksonville, Florida
  - Moffitt McKinley Outpatient Center ( Site 0131), Tampa, Florida
  - Winship Cancer Institute of Emory University ( Site 0046), Atlanta, Georgia
  - Northside Hospital ( Site 0115), Atlanta, Georgia
  - Northwestern Medical Group ( Site 0135), Chicago, Illinois
  - The University of Chicago Medical Center ( Site 0007), Chicago, Illinois
  - Advocate Medical Group-Park Ridge ( Site 0025), Park Ridge, Illinois
  - University of Iowa Hospital and Clinics ( Site 0001), Iowa City, Iowa
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins ( Site 0047), Baltimore, Maryland
  - Massachusetts General Hospital ( Site 0126), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center ( Site 0141), Boston, Massachusetts
  - Dana Farber Cancer Institute ( Site 0124), Boston, Massachusetts
  - Karmanos Cancer Institute ( Site 0111), Detroit, Michigan
  - Mayo Clinic [Rochester, MN] ( Site 0016), Rochester, Minnesota
  - Siteman Cancer Center ( Site 0143), St Louis, Missouri
  - Memorial Sloan Kettering ( Site 0006), Harrison, New York
  - Laura and Isaac Perlmutter Cancer Center ( Site 0137), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0142), New York, New York
  - Mount Sinai Medical Center ( Site 0038), New York, New York
  - University of Rochester ( Site 0019), Rochester, New York
  - The Lindner Center for Research and Education at The Christ Hospital ( Site 0004), Cincinnati, Ohio
  - Stephenson Cancer Center ( Site 0042), Oklahoma City, Oklahoma
  - Oregon Health & Science University ( Site 0032), Portland, Oregon
  - Children's Hospital of Pittsburgh UPMC ( Site 0144), Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Centers ( Site 0043), Pittsburgh, Pennsylvania
  - West Cancer Center - East Campus ( Site 0022), Germantown, Tennessee
  - University of Tennessee Medical Center Knoxville ( Site 0116), Knoxville, Tennessee
  - University of Texas-MD Anderson Cancer Center ( Site 0134), Houston, Texas
  - Inova Schar Cancer Institute ( Site 0014), Fairfax, Virginia
  - VCU Massey Cancer Center ( Site 0008), Richmond, Virginia
  - Seattle Cancer Care Alliance ( Site 0044), Seattle, Washington
  - University of Wisconsin Hospital and Clinics ( Site 0030), Madison, Wisconsin
- Australia (9):
  - Melanoma Institute Australia ( Site 0856), North Sydney, New South Wales
  - Westmead Hospital ( Site 0853), Westmead, New South Wales
  - Cairns Base Hospital ( Site 0859), Cairns, Queensland
  - Tasman Oncology Research Pty Ltd ( Site 0858), Southport, Queensland
  - Princess Alexandra Hospital ( Site 0857), Woolloongabba, Queensland
  - Royal Adelaide Hospital ( Site 0861), Adelaide, South Australia
  - Ashford Cancer Centre Research ( Site 0860), Kurralta Park, South Australia
  - The Alfred Hospital ( Site 0852), Melbourne, Victoria
  - Fiona Stanley Hospital ( Site 0851), Murdoch, Western Australia
- Belgium (6):
  - GZA Sint Augustinus ( Site 0259), Wilrijk - Antwerpen, Antwerpen
  - Institut Jules Bordet ( Site 0254), Brussels, Bruxelles-Capitale, Region de
  - Cliniques Universitaires Saint-Luc ( Site 0251), Brussels, Bruxelles-Capitale, Region de
  - Jessa Ziekenhuis Campus Virga Jesse ( Site 0256), Hasselt, Limburg
  - UZ Gent ( Site 0255), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 0252), Leuven, Vlaams-Brabant
- Brazil (10):
  - Hospital Erasto Gaertner ( Site 0159), Curitiba, Paraná
  - Hospital de Caridade de Ijui ( Site 0156), Ijuí, Rio Grande do Sul
  - Hospital Sao Vicente de Paulo ( Site 0158), Passo Fundo, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da Pucrs ( Site 0154), Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos ( Site 0155), Barretos, São Paulo
  - Hospital de Clinicas de Rio Preto ( Site 0162), Sao Jose Do Rio Preto - SP, São Paulo
  - Instituto Nacional do Cancer II ( Site 0160), Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 0151), São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia ( Site 0161), São Paulo
  - A.C. Camargo Cancer Center ( Site 0164), São Paulo
- Canada (10):
  - Cross Cancer Institute ( Site 0057), Edmonton, Alberta
  - CancerCare Manitoba ( Site 0053), Winnipeg, Manitoba
  - Moncton Hospital - Horizon Health Network ( Site 0055), Moncton, New Brunswick
  - The Ottawa Hospital ( Site 0058), Ottawa, Ontario
  - Sunnybrook Research Institute ( Site 0060), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0059), Toronto, Ontario
  - Hopital Maisonneuve Rosemont ( Site 0056), Montreal, Quebec
  - Jewish General Hospital ( Site 0054), Montreal, Quebec
  - McGill University Health Centre ( Site 0062), Montreal, Quebec
  - CHU de Quebec - Hotel-Dieu de Quebec ( Site 0061), Québec, Quebec
- Chile (6):
  - Fundacion Arturo Lopez Perez FALP ( Site 0200), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0201), Santiago, Region M. de Santiago
  - Sociedad Medica Aren y Bachero Limitada ( Site 0207), Santiago, Region M. de Santiago
  - Instituto Clinico Oncologico del Sur ( Site 0203), Temuco, Región de la Araucanía
  - Oncocentro ( Site 0204), Viña del Mar, Región de Valparaíso
  - Centro Oncologico Antofagasta ( Site 0206), Antofagasta
- France (14):
  - Hopital La Timone ( Site 0302), Marseille, Bouches-du-Rhone
  - CHU Dijon Bourgogne ( Site 0320), Dijon, Cote-d Or
  - CHU de Bordeaux- Hopital Saint Andre ( Site 0304), Bordeaux, Gironde
  - Institut Claudius Regaud IUCT Oncopole ( Site 0306), Toulouse, Haute-Garonne
  - Hopital Ambroise Pare Boulogne ( Site 0316), Boulogne-Billancourt, Hauts-de-Seine
  - CHU Montpellier. ( Site 0312), Montpellier, Herault
  - Centre Eugene Marquis ( Site 0305), Rennes, Ille-et-Vilaine
  - CHU Angers ( Site 0321), Angers, Maine-et-Loire
  - CHU de Reims ( Site 0307), Reims, Marne
  - CHRU Lille - Hopital Claude Huriez ( Site 0301), Lille, Nord
  - C.H.U. Lyon Sud ( Site 0303), Pierre-Bénite, Rhone
  - CHU Amiens Picardie Hopital Nord ( Site 0317), Amiens, Somme
  - Institut Gustave Roussy ( Site 0300), Villejuif, Val-de-Marne
  - Hopital Saint Louis ( Site 0322), Paris
- Germany (11):
  - Universitaetsklinikum in Mannheim ( Site 0351), Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen ( Site 0353), Tübingen, Baden-Wurttemberg
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen ( Site 0357), Munich, Bavaria
  - Klinikum Nuernberg Nord ( Site 0355), Nuremberg, Bavaria
  - Klinikum der Universitaet in Wuerzburg ( Site 0356), Würzburg, Bavaria
  - Elbe Klinikum Buxtehude ( Site 0354), Buxtehude, Lower Saxony
  - Medizinische Hochschule Hannover ( Site 0358), Hanover, Lower Saxony
  - Klinik und Poliklinik fuer Dermatologie Venerologie und Allergologie ( Site 0361), Essen, North Rhine-Westphalia
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel ( Site 0359), Kiel, Schleswig-Holstein
  - SRH Wald-Klinikum Gera GmbH ( Site 0360), Gera, Thuringia
  - Universitaetsklinikum Hamburg Eppendorf (UKE) ( Site 0352), Hamburg
- Israel (7):
  - Soroka Medical Center ( Site 0653), Beersheba, Southern District
  - Sourasky Medical Center ( Site 0656), Tel Aviv, Tell Abib
  - HaEmek Medical Center ( Site 0655), Afula
  - Rambam Medical Center ( Site 0654), Haifa
  - Hadassah Ein Kerem Medical Center ( Site 0651), Jerusalem
  - Chaim Sheba Medical Center. ( Site 0652), Ramat Gan
  - Shamir Medical Center-Assaf Harofeh ( Site 0657), Ẕerifin
- Italy (9):
  - Istituto Scientifico Romagnolo per Studio e Cura Tumori IRST ( Site 0403), Meldola, Forli-Cesena
  - IRCCS Giovanni Paolo II. Ospedale Oncologico ( Site 0406), Bari
  - ASST Papa Giovanni XXIII ( Site 0402), Bergamo
  - IRCCS A.O.U. San Martino - IST ( Site 0404), Genova
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 0408), Milan
  - Istituto Nazionale Tumori Fondazione Pascale ( Site 0400), Napoli
  - IRCCS Istituto Oncologico Veneto ( Site 0407), Padua
  - IDI - Istituto Dermopatico dell'Immacolata ( Site 0405), Roma
  - Azienda Ospedaliero Universitaria Senese ( Site 0401), Siena
- National Cancer Center Hospital ( Site 0910), Tokyo, Japan
- Poland (10):
  - Szpital Kliniczny im. Heliodora Swiecickiego Uniwers Medyczn ( Site 0753), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka ( Site 0769), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Pratia MCM Krakow ( Site 0773), Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 0751), Warsaw, Masovian Voivodeship
  - Instytut Pomnik Centrum Zdrowia Dziecka ( Site 0759), Warsaw, Masovian Voivodeship
  - Kliniczny Szpital Wojewodzki Nr 1 ( Site 0758), Rzeszów, Podkarpackie Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 0770), Gdansk, Pomeranian Voivodeship
  - Beskidzkie Centrum Onkologii im. Jana Pawla II ( Site 0754), Bielsko-Biala, Silesian Voivodeship
  - Uniwersyteckie Centrum Kliniczne Slaskiego Uniwersytetu Medycznego ( Site 0757), Katowice, Silesian Voivodeship
  - LIFTMED ( Site 0765), Rybnik, Silesian Voivodeship
- South Africa (7):
  - Cancer Care Langenhoven Drive Oncology Centre ( Site 0812), Port Elizabeth, Eastern Cape
  - Sandton Oncology Medical Group PTY LTD ( Site 0801), Johannesburg, Gauteng
  - Charlotte Maxeke Johannesburg Academic Hospital ( Site 0811), Parktown, Gauteng
  - Wilgers Oncology Centre ( Site 0806), Pretoria, Gauteng
  - MPOC ( Site 0803), Pretoria, Gauteng
  - Cancercare ( Site 0810), Cape Town, Limpopo
  - Cape Town Oncology Trials Pty Ltd ( Site 0807), Kraaifontein, Western Cape
- Spain (6):
  - Onkologikoa - Instituto Oncologico de San Sebastian ( Site 0457), Donostia / San Sebastian, Gipuzkoa
  - Hospital General Universitario de Valencia ( Site 0451), Valencia, Valenciana, Comunitat
  - Hospital General Universitari Vall d Hebron ( Site 0456), Barcelona
  - Hospital Clinic de Barcelona ( Site 0452), Barcelona
  - Hospital General Universitario Gregorio Maranon ( Site 0454), Madrid
  - Hospital Universitario Virgen Macarena ( Site 0455), Seville
- Switzerland (9):
  - Universitaetsspital Basel ( Site 0554), Basel, Canton of Basel-City
  - Universitaetsspital Bern ( Site 0552), Bern, Canton of Bern
  - Hopitaux Universitaires de Geneve HUG ( Site 0556), Geneva, Canton of Geneva
  - Kantonsspital St. Gallen ( Site 0559), Sankt Gallen, Canton of St. Gallen
  - Centre Hospitalier Universitaire Vaudois ( Site 0553), Lausanne, Canton of Vaud
  - Universitaetsspital Zuerich ( Site 0551), Zurich, Canton of Zurich
  - Oncological Institute of Southern Switzerland ( Site 0557), Bellinzona, Canton Ticino
  - Kantonsspital Graubuenden ( Site 0555), Chur, Kanton Graubünden
  - Hopital du Valais ( Site 0558), Sion, Valais
- United Kingdom (5):
  - Addenbrooke's Hospital in Cambridge ( Site 0600), Cambridge, Cambridgeshire
  - Guy s & St Thomas NHS Foundation Trust ( Site 0601), London, London, City of
  - Royal Marsden Hospital - Fulham Road London ( Site 0613), London, London, City of
  - The Royal Marsden NHS Foundation Trust. ( Site 0612), Sutton, Surrey
  - Christie NHS Foundation Trust ( Site 0604), Manchester

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Luke JJ, Ascierto PA, Khattak MA, de la Cruz Merino L, Del Vecchio M, Rutkowski P, Spagnolo F, Mackiewicz J, Chiarion-Sileni V, Kirkwood JM, Robert C, Grob JJ, de Galitiis F, Schadendorf D, Carlino MS, Wu XL, Fukunaga-Kalabis M, Krepler C, Eggermont AMM, Long GV. Pembrolizumab Versus Placebo as Adjuvant Therapy in Resected Stage IIB or IIC Melanoma: Final Analysis of Distant Metastasis-Free Survival in the Phase III KEYNOTE-716 Study. J Clin Oncol. 2024 May 10;42(14):1619-1624. doi: 10.1200/JCO.23.02355. Epub 2024 Mar 7. PMID 38452313
- [Derived] Luke JJ, Ascierto PA, Khattak MA, Rutkowski P, Del Vecchio M, Spagnolo F, Mackiewicz J, Merino LC, Chiarion-Sileni V, Kirkwood JM, Robert C, Schadendorf D, de Galitiis F, Carlino MS, Dummer R, Mohr P, Odeleye-Ajakaye A, Fukunaga-Kalabis M, Krepler C, Eggermont AMM, Long GV. Pembrolizumab versus placebo as adjuvant therapy in resected stage IIB or IIC melanoma: Long-term follow-up, crossover, and rechallenge with pembrolizumab in the phase III KEYNOTE-716 study. Eur J Cancer. 2025 May 2;220:115381. doi: 10.1016/j.ejca.2025.115381. Epub 2025 Mar 23. PMID 40198940
- [Derived] Wurcel V, Rojas Rojas M, Urrego-Reyes J, Medrano Rivera D, Acevedo R, Jiang R, Jiang S, Zhang S, Caparros A, Krepler C, Fukunaga-Kalabis M, Younan ND, Alexander D, Hughes R, Weston G. Number needed to treat (NNT) with pembrolizumab as an adjuvant therapy in resected patients with high-risk stage II (IIB and IIC) melanoma and its application to cost of preventing an event (COPE) in Mexico. J Med Econ. 2025 Dec;28(1):346-353. doi: 10.1080/13696998.2025.2466365. Epub 2025 Mar 13. PMID 40078077
- [Derived] Schadendorf D, Luke JJ, Ascierto PA, Long GV, Rutkowski P, Khattak A, Del Vecchio M, de la Cruz-Merino L, Mackiewicz J, Sileni VC, Kirkwood JM, Robert C, Grob JJ, Dummer R, Carlino MS, Zhao Y, Kalabis M, Krepler C, Eggermont A, Scolyer RA. Pembrolizumab versus placebo as adjuvant therapy in resected stage IIB or IIC melanoma: Outcomes in histopathologic subgroups from the randomized, double-blind, phase 3 KEYNOTE-716 trial. J Immunother Cancer. 2024 Mar 13;12(3):e007501. doi: 10.1136/jitc-2023-007501. PMID 38485189
- [Derived] Favre-Bulle A, Bencina G, Zhang S, Jiang R, Andritschke D, Bhadhuri A. Cost-effectiveness of pembrolizumab as an adjuvant treatment for patients with resected stage IIB or IIC melanoma in Switzerland. J Med Econ. 2023 Jan-Dec;26(1):283-292. doi: 10.1080/13696998.2023.2174748. PMID 36748342
- [Derived] Long GV, Luke JJ, Khattak MA, de la Cruz Merino L, Del Vecchio M, Rutkowski P, Spagnolo F, Mackiewicz J, Chiarion-Sileni V, Kirkwood JM, Robert C, Grob JJ, de Galitiis F, Schadendorf D, Carlino MS, Mohr P, Dummer R, Gershenwald JE, Yoon CH, Wu XL, Fukunaga-Kalabis M, Krepler C, Eggermont AMM, Ascierto PA; KEYNOTE-716 Investigators. Pembrolizumab versus placebo as adjuvant therapy in resected stage IIB or IIC melanoma (KEYNOTE-716): distant metastasis-free survival results of a multicentre, double-blind, randomised, phase 3 trial. Lancet Oncol. 2022 Nov;23(11):1378-1388. doi: 10.1016/S1470-2045(22)00559-9. Epub 2022 Oct 18. PMID 36265502
- [Derived] Luke JJ, Rutkowski P, Queirolo P, Del Vecchio M, Mackiewicz J, Chiarion-Sileni V, de la Cruz Merino L, Khattak MA, Schadendorf D, Long GV, Ascierto PA, Mandala M, De Galitiis F, Haydon A, Dummer R, Grob JJ, Robert C, Carlino MS, Mohr P, Poklepovic A, Sondak VK, Scolyer RA, Kirkwood JM, Chen K, Diede SJ, Ahsan S, Ibrahim N, Eggermont AMM; KEYNOTE-716 Investigators. Pembrolizumab versus placebo as adjuvant therapy in completely resected stage IIB or IIC melanoma (KEYNOTE-716): a randomised, double-blind, phase 3 trial. Lancet. 2022 Apr 30;399(10336):1718-1729. doi: 10.1016/S0140-6736(22)00562-1. Epub 2022 Apr 1. PMID 35367007
- [Derived] Luke JJ, Ascierto PA, Carlino MS, Gershenwald JE, Grob JJ, Hauschild A, Kirkwood JM, Long GV, Mohr P, Robert C, Ross M, Scolyer RA, Yoon CH, Poklepovic A, Rutkowski P, Anderson JR, Ahsan S, Ibrahim N, M Eggermont AM. KEYNOTE-716: Phase III study of adjuvant pembrolizumab versus placebo in resected high-risk stage II melanoma. Future Oncol. 2020 Jan;16(3):4429-4438. doi: 10.2217/fon-2019-0666. Epub 2019 Dec 24. PMID 31870188
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26208&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, response/progression or adverse events (AEs) during re-challenge/switch-over in Part 2 were not counted towards the recurrence-free survival (RFS) outcome measure or safety outcome measures respectively.
Groups:
- Pembrolizumab: Participants received 200 mg pembrolizumab (2 mg/kg for a maximum of 200 mg in pediatric participants) by intravenous (IV) infusion once every 3 weeks (Q3W; 21-day cycles) for up to 17 cycles (up to ~1 year) in Part 1. Participants who completed the initial treatment of 17 cycles of pembrolizumab and experienced disease recurrence may have been eligible for re-challenge with pembrolizumab at the same dose and schedule of 200 mg Q3W (21-day cycles) for up to 35 cycles (up to ~2 years) in Part 2.
- Placebo: Participants received saline placebo by IV infusion Q3W (21-day cycles) for up to 17 cycles (up to ~1 year) in Part 1. Participants who completed the initial treatment of 17 cycles of placebo and experienced disease recurrence may have been eligible to switch over to pembrolizumab 200 mg Q3W (21-day cycles) for up to 35 cycles (up to ~2 years) in Part 2.
Period: Overall Study
Arm/Group | Pembrolizumab | Placebo
Started | 487 | 489
Treated | 483 | 486
Re-challenged or Switched-over to Pembrolizumab | 1 | 45
Completed | 0 | 0
Not Completed | 487 | 489
Not completed — Ongoing in Study | 460 | 459
Not completed — Withdrawal by Subject | 9 | 10
Not completed — Lost to Follow-up | 1 | 3
Not completed — Death | 17 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Placebo | Total
Number analyzed (Participants) | 487 | 489 | 976
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.0 (12.6) | 59.6 (13.3) | 59.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 200 | 387
  Male | 300 | 289 | 589
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49 | 30 | 79
  Not Hispanic or Latino | 390 | 409 | 799
  Unknown or Not Reported | 48 | 50 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 435 | 439 | 874
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 42 | 45 | 87
Melanoma Primary Tumor (T) Stage [Count of Participants; unit: Participants] — Participants were stratified into T stages of melanoma, as defined by tumor thickness and ulceration, based on the American Joint Committee on Cancer (AJCC) 8th edition. The T stages were defined as follows: T3a: >2.0 - 4.0 mm thickness without ulceration; T3b: >2.0 - 4.0 mm thickness with ulceration; T4a: >4.0 mm without ulceration; T4b: >4.0 mm with ulceration.
  Participants
    T3a | 2 | 0 | 2
    T3b | 200 | 201 | 401
    T4a | 113 | 116 | 229
    T4b | 172 | 172 | 344

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival (RFS)
Description: RFS was defined as the time from randomization to any of the following events: recurrence of melanoma at any site (local, in-transit or regional lymph nodes or distant recurrence) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) or death due to any cause, whichever occurs first. Per protocol, final analysis for this primary outcome measure was performed using the initial pembrolizumab or placebo treatment with a protocol-specified analysis data cut-off date of June-21-2021.
Time Frame: Up to ~32.7 months
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pembrolizumab: Participants received 200 mg pembrolizumab (2 mg/kg for a maximum of 200 mg in pediatric participants) by intravenous (IV) infusion once every 3 weeks (Q3W; 21-day cycles) for up to 17 cycles (up to ~1 year) in Part 1.
- Placebo: Participants received saline placebo by IV infusion Q3W (21-day cycles) for up to 17 cycles (up to ~1 year) in Part 1.
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 487 | 489
Months | NA [NA to NA] — Median, Upper limit and lower limit not reached at the time of data cut-off due to insufficient number of participants with recurrence. | NA [29.9 to NA] — Median and Upper limit not reached at the time of data cut-off due to insufficient number of participants with recurrence.
Statistical Analysis 1: Comparison: Pembrolizumab vs Placebo; Test type: Superiority; p = 0.00046, Log Rank — One-sided p-value based on log-rank test stratified by melanoma T Stage (T3b, T4a, T4b); Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.45 to 0.82] — Hazard Ratio based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by melanoma T Stage (T3b, T4a, T4b)

2. Secondary Outcome: Distant Metastasis-free Survival (DMFS)
Description: DMFS will be defined as the time from randomization to the first diagnosis of a distant metastasis per RECIST 1.1. Distant metastasis will refer to cancer that has spread from the original (primary) tumor and beyond local tissues and lymph nodes to distant organs or distant lymph nodes. DMFS will be reported for randomized participants.
Time Frame: Up to ~9 years
Reporting Status: Not Posted, anticipated posting 2033-10

3. Secondary Outcome: Overall Survival (OS)
Description: OS will be defined as the time from randomization to death due to any cause. OS will be reported for randomized participants.
Time Frame: Up to ~15 years
Reporting Status: Not Posted, anticipated posting 2033-10

4. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Per protocol, analysis for this outcome measure was performed using the initial pembrolizumab or placebo treatment.
Time Frame: Up to ~19.3 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 483 | 486
Participants | 461 | 444
Statistical Analysis 1: Comparison: Pembrolizumab vs Placebo; Test type: Other — Difference in percentage based on Miettinen & Nurminen method; Difference in Percentage = 4.1, 95% CI 2-sided [1.0 to 7.3]

5. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: as for outcome 4
Time Frame: Up to ~19.3 months
Population: All randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 483 | 486
Participants | 84 | 22
Statistical Analysis 1: Comparison: Pembrolizumab vs Placebo; Test type: Other — Difference in percentage based on Miettinen & Nurminen method; Difference in percentage = 12.9, 95% CI 2-sided [9.1 to 16.9]

ADVERSE EVENTS:
Time Frame: All-cause mortality (ACM) : Up to ~32.7 months and safety: Up to ~30.2 months
Description: ACM was analyzed in all randomized participants. Safety was analyzed in all participants who received ≥1 dose of study drug. Per protocol disease progression of cancer was not considered an AE unless related to study drug. Thus MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression", "Disease progression" unrelated to study drug are excluded as AEs. ACM and Safety were analyzed separately in participants who switched over from placebo to pembrolizumab.
Groups:
- Placebo Switched Over to Pembrolizumab: Participants who received the initial treatment of saline placebo by IV infusion Q3W (21-day cycles) for up to 17 cycles (up to ~1 year) in Part 1 and experienced disease recurrence may have been eligible to switch over to pembrolizumab 200 mg Q3W (21-day cycles) for up to 35 cycles (up to ~2 years) in Part 2.
Arm/Group | Pembrolizumab | Placebo | Placebo Switched Over to Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 17/487 | 18/489 | 3/45
Serious Adverse Events (participants affected / at risk) | 101/483 | 91/486 | 6/45
Other Adverse Events (participants affected / at risk) | 417/483 | 364/486 | 26/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=483) | Placebo (N=486) | Placebo Switched Over to Pembrolizumab (N=45)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (5) | 1 (1) | 0 (0)
Autoimmune myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 4 (4) | 0 (0) | 0 (0)
Endocrine disorder (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Macular detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion site urticaria (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 3 (3) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Abscess soft tissue (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Cellulitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected seroma (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Ultrasound bladder abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (23) | 24 (53) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 5 (6) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 6 (6) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Mucinous adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (11) | 14 (18) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Myelitis transverse (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgic amyotrophy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=483) | Placebo (N=486) | Placebo Switched Over to Pembrolizumab (N=45)
Hyperthyroidism (Endocrine disorders) | 50 (50) | 3 (4) | 4 (4)
Hypothyroidism (Endocrine disorders) | 82 (82) | 16 (16) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 30 (37) | 24 (29) | 2 (3)
Constipation (Gastrointestinal disorders) | 40 (46) | 40 (45) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 134 (222) | 96 (176) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 31 (33) | 9 (10) | 3 (3)
Nausea (Gastrointestinal disorders) | 66 (100) | 56 (90) | 0 (0)
Vomiting (Gastrointestinal disorders) | 31 (40) | 15 (17) | 1 (1)
Asthenia (General disorders) | 54 (75) | 53 (80) | 3 (3)
Fatigue (General disorders) | 140 (161) | 122 (137) | 2 (2)
Oedema peripheral (General disorders) | 28 (35) | 22 (23) | 0 (0)
Pyrexia (General disorders) | 31 (32) | 26 (26) | 3 (3)
Nasopharyngitis (Infections and infestations) | 22 (27) | 29 (35) | 2 (2)
Alanine aminotransferase increased (Investigations) | 55 (63) | 29 (38) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 36 (42) | 19 (22) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 26 (31) | 12 (15) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (16) | 28 (36) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 113 (155) | 83 (107) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 40 (44) | 37 (38) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 50 (56) | 28 (29) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 (29) | 28 (31) | 1 (2)
Dizziness (Nervous system disorders) | 32 (38) | 27 (29) | 3 (3)
Headache (Nervous system disorders) | 81 (102) | 55 (70) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 56 (65) | 57 (65) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 (22) | 25 (32) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 131 (177) | 61 (78) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 89 (116) | 41 (52) | 2 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 40 (52) | 9 (13) | 0 (0)
Hypertension (Vascular disorders) | 40 (49) | 43 (61) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT03553836/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT03553836/SAP_001.pdf